

## **Data Analysis Plan**

**Project Title**: Adapting a Peer-Delivered Behavioral Activation Intervention to Improve Adherence to MAT among Low-Income, Minority Individuals with OUD

Principal Investigator: Jessica F. Magidson, PhD

**Grant:** R61AT010799

Version Date: 21 September 2022

Primary Outcomes

Descriptive statistics were used to characterize the sample, including implementation outcomes. We defined benchmark milestones *a priori* for successful implementation:  $\geq$ 75% of patients participating in the first *Peer Activate* session (feasibility);  $\geq$ 75% of patients completing  $\geq$ 75% of the core *Peer Activate* sessions (acceptability); and PRS fidelity  $\geq$ 75% as rated by an independent coder. Methadone retention was examined using descriptive and inferential analyses.

## **Implementation Outcomes**

**Feasibility** measured using qualitative feedback and quantitatively as the % of patients who agree to participate in the intervention.

Quantitatively, ≥75% of patients agreeing to participate in the intervention will be considered feasible.

Qualitatively, feasibility as defined by Proctor's model and coded by two independent coders.

<u>Acceptability</u> measured using qualitative feedback and quantitatively as the % of patients enrolled who attend ≥75% of the core sessions.

Quantitatively, ≥75% of patients attending ≥75% of the core sessions will be considered acceptable.

Qualitatively, acceptability as defined by Proctor's model and coded by two independent coders.

<u>Fidelity</u> measured based on peer adherence to the intervention manual. A random selection of 20% of sessions were rated for fidelity, and ≥75% of session components delivered as intended will be considered the threshold for fidelity.